CLINICAL TRIAL: NCT05393349
Title: 'Home Sweet Home' Programme: Empowering the Patient and Caregiver for Early and Safe Discharge of Patients With Geriatric Hip Fractures
Brief Title: Geriatric Hip Fractures Caregiver Programme
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wong Tak-Man, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 19-574
Record Dates: First submitted 2022-04-26; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Geriatric Hip Fracture
Keywords: Empowerment; Caregiver; Geriatric Hip Fractures; Functional outcomes
MeSH Terms: conditions — Empowerment | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Empowering the patient and caregiver for early and safe discharge of patients with geriatric hip fractures
- Standard Group (No Intervention)

INTERVENTIONS:
Behavioral: Empowering the patient and caregiver for early and safe discharge of patients with geriatric hip fractures — Orthopaedic surgeon, geriatrician, physiotherapists, occupational therapists, and nurses will make videos (each 3-5 minutes long) which are available to the patients and caregivers during both the hospitalization period and after discharge. They will complement the therapists' training sessions and allow revision of the contents by the patients and caregivers anytime. The patients and caregivers will be asked to complete an assessment after they view the videos to reinforce the knowledge they learn in the videos. Caregivers can be patient's relatives, friends or domestic helper who can commit to visiting the patient at least two days per week during the early discharge period.
  Arms: Intervention Group

SUMMARY:
Objective:

To study whether fracture hip patients can be benefited from the empowerment program

Hypothesis to be tested Primary hypothesis: empowerment program can improve the patient's functional recovery.

Secondary hypothesis: the program can improve readmission rate, length of stay, and secondary fracture.

Design and subjects This is a prospective randomised controlled trial and subjects are fracture hip patients

Instruments Ipads are needed to show the videos of the rehabilitation program

Interventions

The empowerment program consists of three main areas which directly correspond to the contents that the patients and caregivers expressed as most needed in interviews conducted by the investigators during hip fracture patients' follow up:

* Knowledge of the disease
* Confidence and skills in self-care management
* Support in the post-discharge period

Main outcome measures

Primary outcomes:

Functional scores (Modified Barthel Index and EQ-5D-5L) at the first follow-up visit (3 months postop).

Timed-up-and-go test at follow-up at 6 months and 1 year.

Secondary outcome:

Cumulative readmission rates at 1 month, 6 months, and 1 year The length of stay in the convalescent hospital Subsequent injury with fractures within 1 year

Data analysis Chi-square test is used for categorical variables. For continuous variables, the normal distribution is determined by the Kolmogorov-Smirnov test. Independent t-test is used for comparing average values of normally distributed continuous variables, while the Wilcoxon rank sum test is used for comparing median values of abnormally distributed variables.

Binary logistic regression is used to determine predictive factors for outcomes. Multivariate analysis is performed to verify independent predictive factors for outcomes.

Expected results Fracture hip patients can be benefited from the empowerment program.

DETAILED DESCRIPTION:
Introduction:

Health care consequences of hip fracture The global incidence of geriatric hip fractures is projected to increase by more than 250% in the next twenty-five years. Local data showed that there was a steady increase from 3500 to more than 4500 hip fractures per year from 2000 to 2011. Nevertheless, the consequence of hip fractures is serious and costly. Ten percent of patients have a contralateral hip fracture, 30% of the patients are readmitted for other acute reasons, 25% need long-term care, 10-25% die within 1 year and almost 50% have residual functional disabilities.

Geriatric hip fracture clinical pathway decreased preoperative length of stay Since 2006, the geriatric hip fracture clinical pathway (GFH) has been implemented in the Hong Kong West Cluster. The implementation of GFH resulted in a decreased preoperative length of stay, decreased surgical site infection, decreased pressure sore, and decreased 30-day and 12-month mortality rate.

High dependency of patients upon discharge:

However, according to our data, a significant number of patients still required an extended length of stay, which is defined as more than 28 days in a rehabilitation hospital. More than 60% of the patients were discharged home, however, 39% and 51% of the patients had severe and moderate dependency respectively upon discharge from the rehabilitation hospital (Modified Barthel Index 0-60 and 61-90 respectively). Current training provided to those patients and their caregivers was brief and inadequate. The lack of a trained caregiver affects the decision to return home and patients may need settlement in nursing homes. Moreover, 12% had readmission within 28 days of discharge, with repeated falls accounting for the majority.

The patients were referred to a geriatric day hospital after discharge from the convalescent hospital. However, the waiting time for geriatric day hospital was 2 months. During this interval, the patients were discharged home and taken care of by the caregivers. The caregivers were unsupported and inadequately trained for the job.

Patient and caregiver empowerment for hip fracture patients in Hong Kong:

Patient empowerment has been used in patients with stroke and other geriatric conditions. There are only scarce studies focussing on geriatric hip fractures which required special care in terms of ambulation, transfers, and activities of daily living training. So far prospective randomized studies are lacking. A previous study showed patient empowerment resulted in a shortened length of stay and earlier return to previous living by comparing two hospitals.

In Hong Kong, the elderly hip fracture patients returning home are often taken care of by domestic helpers or family members. Caring for older patients after hospital discharge is challenging and many of their caregivers lack the confidence to do so. Hence, we opine that caregivers need special attention as well. Another study also studied the caregivers' burden of hip fracture patients in Taiwan. The caregivers experienced moderate burdens. Caregivers who could not access other resources for help experienced a higher burden.

There has been an increasing trend for patient and caregiver empowerment programs. A study done by Hendrix (2013) investigated the effects of an individualized caregiver training program on self-efficacy in-home care and symptom management. Results revealed a significant increase in self-efficacy after the training in the treatment group, however, their study focused on cancer patients only. Another study done by Coleman in the year 2004 tested whether an intervention designed to encourage older patients and their caregivers to assert a more active role during discharge could result in decreased rehospitalization rates. He showed the adjusted odds ratio comparing rehospitalization of intervention subjects with that of controls was 0.52 at 30 days, 0.43 at 90 days, and 0.57 at 180 days. Intervention patients reported high levels of confidence in obtaining essential information for managing their condition, communicating with members of the healthcare team, and understanding their medication regimen. Their patient population is heterogeneous and includes various medical and orthopaedic patients.

Most studies on patient and caregiver empowerment had shown positive results. The proposed study focuses on empowering hip fracture patients and their caregivers in all aspects in terms of ambulation, transfers, and activities of daily living training. The impact of empowerment on hip fracture patients and their caregivers has not been studied in Hong Kong and the aim of the project is to investigate if those fracture hip patients can be benefited from the empowerment program in terms of functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65
2. Acute intracapsular or extracapsular proximal femur fracture
3. Surgical treatment: Hemiarthroplasty or reduction-internal fixation
4. Availability of caregiver

Exclusion Criteria:

1. No caregiver support
2. Non-operative treatment
3. Pathological fracture
4. Multiple fractures
5. Patient discharged directly from the acute hospital without convalescence 6. Premorbid bedbound/chairbound status

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional scores | First follow up visit (3 months postop)
  Modified Barthel Index
Functional scores | First follow up visit (3 months postop)
  EQ-5D-5L
Walking function | 6 months
  Timed-up-and-go test
Walking function | 1 year
  Timed-up-and-go test

SECONDARY OUTCOMES:
Cumulative readmission rates | 1 month after hip surgery
Cumulative readmission rates | 6 months after hip surgery
Cumulative readmission rates | 2 years after hip surgery
The length of stay in convalescent hospital | Up to discharge back to home
Number of subsequent injury with fractures | within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tak Man Wong, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided